CLINICAL TRIAL: NCT06437704
Title: The Effects of Brain Training Games on Cognitive Function and Quality of Life Among Older Adults With Mild Cognitive Impairment
Brief Title: Effects of Brain Training Games on Cognitive Function and Quality of Life in MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lylas Ali
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Aging; Quality of life; Brain training games
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Brain training game (Lumosity)
  Interventions: Other: Brain training game Lumosity
- Control (Active Comparator): Simulation game (Simcity buildit)
  Interventions: Other: Simulation game simcity buildit

INTERVENTIONS:
Other: Brain training game Lumosity — . Group A, the experimental group will be trained using five selected games i.e. Speed Match, Memory Matrix, Tidal treasure, Ebb and Flow and Lost in Migration from Lumosity for a period of 30 sessions , 30 min/ day over the span of 6 weeks.
  Arms: Experimental
Other: Simulation game simcity buildit — Group B, the active control will be trained for the same number of sessions using a simulation game, SimCity Build it, for a period of 30 sessions , 30 min/ day over the span of 6 weeks.
  Arms: Control

SUMMARY:
The study aims to determine the effects of brain training games on cognitive function and Quality of life among older adults with MCI.

DETAILED DESCRIPTION:
The study aims to determine the effects of brain training games on cognitive function and Quality of life among older adults with MCI.This study will assess the efficacy of Brain training games. Lumosity on the cognitive function and Quality of life among older adults with MCI .Beyond cognitive rehabilitation, this intervention holds promise as a cost-effective approach to delay, maintain, or even improve cognitive decline associated with the aging process.

ELIGIBILITY:
Inclusion Criteria:

* Older adults of age >50 years and above
* Both male and female
* Education level matriculation at least
* Mild cognitive impairment ( MOCA score of 18-25)
* Active independent individuals with normal hearing and normal or corrected-to-normal vision.

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Diagnosed case of dementia, depression or other mental issues.
* Current plans to move to another city.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-10-16 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale | 6 weeks
  Brief cognitive function assessment is done using MoCA Questionnaire which consist of 12 items, that is to say visuospatial, executive functioning, short-term memory, attention or concentration, working memory, language, and lastly orientation. The total score of this Questionnaire is 30. As per grading system, the score of 26 to 30 represent normal cognition, score of 18 to 25 denotes mild cognitive impairment and score of 10-17 signifies moderate cognitive impairment. Lastly, score of less than 10 embodies severe cognitive impairment. The inter-rater reliability or ICC value is 0.96 (95% CI: 0.91-0.98). Cronbach's alpha is 0.79 and AUC of 0.89 (95% CI: 0.83-0.95).
Trail Making Test A and B | 6 weeks
  Trail making test is a brief paper and pencil test used to screen for any cognitive impairment with the test scored by how long does it takes for a person to complete it. In part A of the test, the patient draw lines to join numbered circles from 1-to 25, connecting them in ascending order. The average score for completing this test is 29 seconds, whereas the rule of thumb suggests a typical score of 90 seconds. A score of greater than 78 seconds indicates deficiency. In part B of the test, the patient connect the circles alternating between numbers from 1 to 13 and letters from A to L. The average score is 75 seconds, with score of greater than 273 seconds representing deficiency. The rule of thumb for this test is a typical score of 3 minutes. The retest reliability for part A is between 0.76 and 0.89 and for part B it lies between 0.86 and 0.94. The Cronbach's alpha for this neuropsychological test is 0.90.
World Health Organization Quality of Life Brief Version (WHO-QOL BREF) Questionnaire: | 6 weeks
  WHO-QOL BREIF questionnaire is a 26 items tool for measuring quality of life. It address four domains of quality of life which includes physical health comprising of 7 items, psychological health having 6 items, social relationships 3 items, and environmental health encompassing 8 items; it also contains QOL and general health items. Each item in the questionnaire is scored on a 5 point ordinal scale; from 1 to 5.The scores are then transformed linearly to a 0 to 100 scale where 0 score represents the worst of health and maximum score of 100 indicates best possible state of health. The Cronbach's alpha coefficient for this questionnaire is 0.86 and the ICC value is 0.74. The CVI score is within the range of 0.78 to 1.00
International Physical Activity Questionnaire (IPAQ); | 6 weeks
  IPAQ is a self-reported tool for the assessment of level of physical activity. It evaluates the duration of physical activity in the last 7 days in the domains of job related physical activity, transportation , house chores and house maintenance, caring for family, recreational activities, sport, and leisure-time physical activity as well as time spent sitting. The score is recorded in the form of MET minutes. The total minutes per week spent on each activity type, that is walking (3.3 METs), doing moderate (4.0 METs) or vigorous physical activity (8.0 METs) are calculated and converted into MET-minutes. The sum of total MET-minutes for each activity determine the level of total physical activity. The questionnaire has an excellent test-retest reliability for physical activity (ICC = 0.84-1.00) as well as an exceptional concurrent validity: ρ = 0.71

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Riphah International University, Gulberg Green Campus, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No